CLINICAL TRIAL: NCT05260294
Title: Identification of Epidural Space: A Comparison Study Between Contrast Spread and Loss of Resistance Techniques
Brief Title: A Comparison Study Between Contrast Spread and Loss of Resistance Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakov Perper, MD (Other)
Responsible Party: Sponsor-Investigator, Yakov Perper, MD, Director of Astoria Pain Management PLLC, Principal Investigator, Astoria Pain Management
Organization: Astoria Pain Management (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-06-002
Record Dates: First submitted 2022-02-02; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Cervical Radiculopathy; Neck Pain; Disc Prolapse With Radiculopathy
Keywords: Fluoroscopy only; cervical epidural steroid injection; contrast spread technique; loss of resistance technique; epidural space identification
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups of 20 each and underwent CESI with either an 18G or a 25G Tuohy needle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18 Gauge Tuohy group (Active Comparator): In the 18G group, all CESIs were performed utilizing the fluoroscopy only method when the needle was navigated from the skin toward the epidural space under contralateral oblique fluoroscopy, and the contrast spread technique was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK).
  Interventions: Procedure: Epidural space identification with cervical epidural steroid injection employing CST and LORT.
- 25 Gauge Tuohy group (Active Comparator): In the 25G group, all CESIs were performed utilizing the fluoroscopy only method when the needle was navigated from the skin toward the epidural space under contralateral oblique fluoroscopy, and the contrast spread technique was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK).
  Interventions: Procedure: Epidural space identification with cervical epidural steroid injection employing CST and LORT.

INTERVENTIONS:
Procedure: Epidural space identification with cervical epidural steroid injection employing CST and LORT. — Cervical epidural procedure and epidural space recognition were performed utilizing the fluoroscopy only method. With this technique, needle navigation from the skin toward the epidural space is performed under contralateral oblique fluoroscopy. With the needle at the ventral interlaminar line, the contrast spread technique was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK). Subsequently, accompanied by the radiology assistant, I observed the Epidrum for 30 seconds or more; if the Epidrum deflated, thus confirming LOR, the result was positive. However, if the device remained inflated, the result was reported as negative. The collected data was then analyzed.

SUMMARY:
Early epidural space identification is critical to the efficacy and safety of cervical epidural steroid injections (CESI) [1]. Currently, the accepted method for epidural space recognition is the loss of resistance technique (LORT). I perform CESIs with fluoroscopy only [2]. I hypothesized that the contrast spread technique (CST) might recognize epidural space concurrently with or sooner than LORT. I also suggested that smaller needles might be employed with CST but not with LORT. To test my hypotheses, I conducted a comparison study.

DETAILED DESCRIPTION:
The study participants were patients of Astoria Pain Management, New York, USA (age 28-72 years) with a clinical diagnosis of cervical radiculitis. The Canadian SHIELD Ethics Review Board approved this study (July 18, 2019. REB tracking number: 19-06-002), conducted from August 19, 2019, to October 8, 2019. There was no funding for this study. Patients were eligible for the study if they met the criteria for cervical ESI, which included clinical and recent MRI findings confirming the diagnosis of cervical radiculitis and inadequate pain relief with conservative care for more than 3 months. Other criteria were if the procedure was covered by medical insurance, and if they signed informed consent. Patients were excluded from the study if they were taking anticoagulants or had serious comorbidities such as congestive heart failure.

The patients were divided into two groups of 20 each and underwent CESI with either an 18G or a 25G Tuohy needle. The skin was anesthetized with 1% lidocaine in the 18G group but not in the 25G group. All cervical epidurals were performed utilizing the fluoroscopy only method when the needle was navigated from the skin toward the epidural space under contralateral oblique fluoroscopy [3], and the contrast spread technique [4,5] was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK). I utilized the Epidrum device as I consider it a more objective and reproducible method for epidural space identification independent of the provider's skill with the LORT, and because its success rate is comparable to the results attained by trained anesthesiologists employing the LOR syringe [6, 7, 8]. Subsequently, accompanied by the radiology assistant, I observed the Epidrum for 30 seconds or more; if the Epidrum deflated, the result was positive. However, if the device remained inflated, the result was reported as negative. The collected data was then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and recent MRI findings confirming the diagnosis of cervical radiculitis
* Inadequate pain relief with conservative care for more than 3 months
* Signed informed consent
* The procedure was covered by medical insurance

Exclusion Criteria:

* Bleeding disorder or anticoagulants therapy
* Serious comorbidities such as congestive heart failure
* Pregnancy
* Uncontrolled diabetes mellitus
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Confirmation of the LOR with epidurally located 18G Tuohy needle by the Epidrum device. | 30 seconds
  Cervical epidural procedure and epidural space recognition were performed utilizing the fluoroscopy only method. With this technique, needle navigation from the skin toward the epidural space is performed under contralateral oblique fluoroscopy. With the needle at the ventral interlaminar line, the contrast spread technique was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK). Subsequently, accompanied by the radiology assistant, I observed the Epidrum for 30 seconds or more; if the Epidrum deflated, thus confirming LOR, the result was positive. However, if the device remained inflated, the result was reported as negative.
Confirmation of the LOR with epidurally located 25G Tuohy needle by the Epidrum device. | 30 seconds
  Cervical epidural procedure and epidural space recognition were performed utilizing the fluoroscopy only method. With this technique, needle navigation from the skin toward the epidural space is performed under contralateral oblique fluoroscopy. With the needle at the ventral interlaminar line, the contrast spread technique was employed for epidural space identification. After radiological confirmation of the epidural spread, LOR was tested using an Epidrum® device (Exmoor Innovations Ltd., Somerset, UK). Subsequently, accompanied by the radiology assistant, I observed the Epidrum for 30 seconds or more; if the Epidrum deflated, thus confirming LOR, the result was positive. However, if the device remained inflated, the result was reported as negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Astoria Pain Management, Astoria, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoffmann VL, Vercauteren MP, Vreugde JP, Hans GH, Coppejans HC, Adriaensen HA. Posterior epidural space depth: safety of the loss of resistance and hanging drop techniques. Br J Anaesth. 1999 Nov;83(5):807-9. doi: 10.1093/bja/83.5.807. PMID 10690148
- [Result] Doan L, Patel H, Aronova Y, Gharibo C. Variations in Interlaminar Epidural Steroid Injection Practice Patterns by Interventional Pain Management Physicians in the United States. Pain Physician. 2018 Sep;21(5):E493-E499. PMID 30282397
- [Result] Furman MB, Jasper NR, Lin HW. Fluoroscopic contralateral oblique view in interlaminar interventions: a technical note. Pain Med. 2012 Nov;13(11):1389-96. doi: 10.1111/j.1526-4637.2012.01484.x. Epub 2012 Sep 19. PMID 22994264
- [Result] Perper Y. Contrast spread technique. Pain Med. 2015 Apr;16(4):827-8. doi: 10.1111/pme.12650. Epub 2015 Feb 4. No abstract available. PMID 25651004
- [Result] Perper Y. Contrast Spread Technique: Evolution. Pain Med. 2016 Jul;17(7):1385-1386. doi: 10.1093/pm/pnv100. Epub 2016 Feb 5. No abstract available. PMID 26849949
- [Result] Kartal S, Kosem B, Kilinc H, Kosker H, Karabayirli S, Cimen NK, Demircioglu RI. Comparison of Epidrum, Epi-Jet, and Loss of Resistance syringe techniques for identifying the epidural space in obstetric patients. Niger J Clin Pract. 2017 Aug;20(8):992-997. doi: 10.4103/1119-3077.214366. PMID 28891544
- [Result] Kim SW, Kim YM, Kim SH, Chung MH, Choi YR, Choi EM. Comparison of loss of resistance technique between Epidrum(R) and conventional method for identifying the epidural space. Korean J Anesthesiol. 2012 Apr;62(4):322-6. doi: 10.4097/kjae.2012.62.4.322. Epub 2012 Apr 23. PMID 22558497
- [Result] Sawada A, Kii N, Yoshikawa Y, Yamakage M. Epidrum((R)): a new device to identify the epidural space with an epidural Tuohy needle. J Anesth. 2012 Apr;26(2):292-5. doi: 10.1007/s00540-011-1278-1. Epub 2011 Nov 13. PMID 22081113
- [Derived] Perper Y. Identification of cervical epidural space: A comparison study between contrast spread and loss of resistance techniques. Front Pain Res (Lausanne). 2022 Dec 20;3:1000209. doi: 10.3389/fpain.2022.1000209. eCollection 2022. PMID 36618582

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT05260294/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT05260294/ICF_001.pdf